CLINICAL TRIAL: NCT05103358
Title: A Phase 2 Multi-center Open-label Basket Trial of Nab-sirolimus for Adult and Adolescent Patients With Malignant Solid Tumors Harboring Pathogenic Inactivating Alterations in TSC1 or TSC2 Genes.
Brief Title: Phase 2 Basket Trial of Nab-sirolimus in Patients With Malignant Solid Tumors With Pathogenic Alterations in TSC1/TSC2 Genes (PRECISION 1)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSC-007
Record Dates: First submitted 2021-10-22; First posted 2021-11-02 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Tumor; Tumor, Solid; Metastasis; Metastatic Cancer; Cancer; Cancer Metastatic; Tumors; Neoplasms; Neoplasm Metastasis; Solid Tumor; Advanced Solid Tumor; Advanced Cancer; Malignant Solid Tumor; Malignant Solid Neoplasm; Malignant Neoplasm; Malignant Tumor; TSC; TSC1; TSC2; Metastatic Solid Tumor; Metastatic Neoplasm
Keywords: TSC1 gene; TSC2 gene; Tissue agnostic; Basket; nab-sirolimus; mTOR inhibitor; nanoparticle albumin bound; mammalian target of rapamycin; mechanistic target of rapamycin; tumor profile; tuberous sclerosis complex 1; tuberous sclerosis complex 2; mTOR; sirolimus; TSC1; TSC2; ABI-009; FYARRO; Precision; Precision 1; Pathogenic alterations; Pathogenic mutations; Inactivating mutations
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Tuberous Sclerosis 1; Tuberous Sclerosis 2; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pathogenic inactivating TSC1 alterations (Experimental): Patients with pathogenic inactivating TSC1 alterations.
  Interventions: Drug: nab-sirolimus
- Arm B: Pathogenic inactivating TSC2 alterations (Experimental): Patients with pathogenic inactivating TSC2 alterations.
  Interventions: Drug: nab-sirolimus

INTERVENTIONS:
Drug: nab-sirolimus — Prospective phase 2, open-label, multi-institutional basket trial to determine the efficacy and safety of nab-sirolimus administered by IV infusion to patients
  Other Names: ABI-009

SUMMARY:
A Phase 2 multi-center open-label basket trial of nab-sirolimus for adult and adolescent patients with malignant solid tumors harboring pathogenic inactivating alterations in TSC1 or TSC2 genes

DETAILED DESCRIPTION:
Study TSC-007 is a prospective phase 2, open-label, multi-institutional basket trial to determine the efficacy and safety profile of nab-sirolimus administered to patients with malignant solid tumors harboring pathogenic inactivating alterations in TSC1 or TSC2 genes. Patients will be treated with single agent IV nab-sirolimus until disease progression, or unacceptable toxicity, or until in the opinion of the investigator the patient is no longer benefiting from therapy, or at patient discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a malignant solid tumor with a pathogenic inactivating TSC1 or TSC2 alteration. Genetic alterations should be identified using NGS in tumor tissue or liquid biopsy).

   • Patients will be enrolled after the central evaluation of NGS report confirms eligibility.
2. Patients must have solid tumors that are metastatic or locally advanced where surgical resection is not an option or likely to result in severe morbidity.
3. Patients must have received all standard therapies appropriate for their tumor type and stage of disease or, in the opinion of the Investigator, the patient would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy, or the patient has no satisfactory alternative treatments.
4. Patients must have 1 or more measurable target lesions by computed tomography (CT) scan or magnetic resonance imaging (MRI) (RECIST v1.1).
5. Age: 12 years or older.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 or Karnofsky Performance Status (KPS) ≥80 or Lansky play-performance scale for pediatric patients ≥80.
7. Adequate liver function:

   1. Total bilirubin ≤1.5 × upper limit of normal (ULN) (unless due to Gilbert's syndrome, then ≤3 × ULN)
   2. Aspartate aminotransferase (AST) ≤2.5 × ULN (≤5 × ULN if attributable to liver metastases)
8. Adequate renal function: creatinine clearance ≥30 mL/min, Cockcroft-Gault CCr = ((140-age) × weight[kg]) / (72 × SCr[mL/min]) × 0.85, if female
9. Adequate hematologic parameters:

   1. Absolute neutrophil count (ANC) ≥1.0 × 109/L (growth factor support allowed)
   2. Platelet count ≥100,000/mm3 (100 × 109/L) (transfusion and/or growth factor support allowed)
   3. Hemoglobin ≥8.0 g/dL (transfusion and/or growth factor support allowed)
10. Fasting serum triglyceride must be ≤300 mg/dL; fasting serum cholesterol must be ≤350 mg/dL.
11. Minimum of 4 weeks since any major surgery, completion of radiation, or completion of prior systemic anticancer therapy, or at least 5 half-lives if the prior therapy is a single agent small-molecule therapeutic, and adequately recovered from the acute toxicities of any prior therapy, including neuropathy, to Grade ≤1.
12. Male or non-pregnant and non-breastfeeding female:

    1. Females of childbearing potential must agree to use effective contraception or abstinence without interruption from 28 days prior to starting investigational product (IP) throughout 3 months after last dose of IP and have a negative serum pregnancy test (beta human chorionic gonadotropin, β-hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. A second form of birth control is required even if she has had a tubal ligation.
    2. Male patients must agree not to donate sperm and must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after last dose of IP. A second form of birth control is required even if he has undergone a successful vasectomy.
13. The patient or the patient's parent(s) or legal guardian(s) understand(s) and sign(s) the informed consent.
14. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Prior treatment with an mTOR inhibitor, including nab-sirolimus.
2. Severe (Grade ≥3) ongoing infection requiring parenteral or oral anti-infective treatment, either ongoing or completed ≤7 days prior to enrollment.
3. Patients with primary brain tumors or PEComa.
4. Patients who have any severe and/or uncontrolled medical or psychiatric conditions or other conditions that could affect their participation including:

   1. Patients with meningeal carcinomatosis, leptomeningeal carcinomatosis, spinal cord compression, untreated brain metastases or symptomatic or unstable brain metastases. Note: Patients with stable brain metastases (defined as asymptomatic or no requirement for high-dose [defined as dexamethasone 10 mg daily or higher] or increasing dose of systemic corticosteroids) and without imminent need of radiation therapy are eligible. If applicable, patients must have completed brain radiation therapy and recovered adequately from any associated toxicity and/or complications prior to eligibility assessment. For patients who have received prior radiation therapy, post-treatment MRI scan should show no increase in brain lesion size/volume.
   2. Unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association, NYHA class III or IV), myocardial infarction ≤6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
   3. Pre-existing severely impaired lung function. If a patient has a pre-existing pulmonary condition, eligible patients should have a spirometry and diffusing capacity for carbon monoxide (DLCO) that is >50% of the normal predicted value and/or O2 saturation that is >88% at rest on room air (Note: spirometry and pulmonary function tests [PFTs] not required to be performed unless clinically indicated).
   4. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy.
   5. A history of malignancies other than the one under treatment unless the patient is disease-free for more than 5 years from diagnosis. Note, controlled non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer, certain low grade hematologic malignancies (eg CLL, follicular lymphoma, etc), or other adequately treated carcinoma-in-situ may be eligible, after discussion with the medical monitor.
   6. Uncontrolled hypertension (systolic blood pressure ≥160 mm-Hg and/or diastolic blood pressure ≥100 mm Hg).
   7. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
   8. Individuals with known human immunodeficiency virus (HIV) infection are excluded from this study as combination antiretroviral therapy could potentially result in significant pharmacokinetic interactions. In addition, these individuals are at increased risk of serious infections due to the immunosuppressive effects of mTOR inhibition.
   9. Active Hepatitis B or Hepatitis C, with detectable viral load.
5. Regarding concomitant medications with significant CYP3A4 and P-gp interactions, discontinuation of strong inhibitors (eg, ketoconazole, itraconazole, voriconazole, erythromycin, clarithromycin, telithromycin, and others), strong inducers (eg, rifampin, rifabutin), and known CYP3A4 substrates with a narrow therapeutic window (eg, fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, or terfenadine) is required at least 5 half lives prior to receiving the first dose of nab-sirolimus, whichever is longer.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 9 months
  ORR based on the proportion of patients with best overall response (BOR) of confirmed partial response (PR) or complete response (CR) from the time of study treatment initiation until disease progression as determined by IRR using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | 9 months
  Determined for patients with BOR of confirmed CR or PR (by IRR)
Disease control rate | 9 months
  BOR of confirmed CR or PR (either of any duration) or stable disease (SD) following study treatment initiation (by IRR)
Time to response | 9 months
  Time from first dose of study drug to initial measurement of CR or PR, where CR or PR is subsequently confirmed
Progression-free survival | 9 months
  Number of months from study treatment initiation to the date of disease progression (by IRR) or death due to any cause
Overall survival | 24 months
  Number of months from study treatment initiation to the date of death due to any cause
Patient-reported outcome | 9 months
  Changes from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire v3.0 (EORTC-QOQ-C30) scores
Incidence and severity of treatment-emergent and treatment-related adverse events (AEs) | 9 months
  Incidence and severity of treatment-emergent and treatment-related AEs as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (159):
- United States (152):
  - Alabama Oncology, Birmingham, Alabama
  - Southern Cancer Center, Mobile, Alabama
  - Arizona Oncology Associates, Goodyear, Arizona
  - Honor Health, Phoenix, Arizona
  - Arizona Oncology Associates, Prescott Valley, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Nextgen Oncology, Beverly Hills, California
  - City of Hope, Duarte, California
  - Providence Medical Foundation (Fullerton), Fullerton, California
  - MemorialCare, Long Beach, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Providence Medical Foundation (Napa), Napa, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sharp HealthCare, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Stanford Cancer Center, Stanford, California
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers (Williams St), Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Hartford Healthcare, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - Florida Cancer Specialists - North Division, Altamonte Springs, Florida
  - Florida Cancer Specialists - South Division, Bonita Springs, Florida
  - Florida Cancer Specialists - South Division, Bradenton, Florida
  - Florida Cancer Specialists - North Division, Brandon, Florida
  - Florida Cancer Specialists - South Division, Cape Coral, Florida
  - Florida Cancer Specialists - North Division, Clearwater, Florida
  - Cancer Specialist - East, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists South Division, Fort Myers, Florida
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North Division, Gainesville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - The Oncology Institute of Hope and Innovation, Lakeland, Florida
  - TOI Florida, Lakeland, Florida
  - Florida Cancer Specialists - North Division, Largo, Florida
  - Florida Cancer Specialists - North Division, Lecanto, Florida
  - Florida Cancer Specialists - South Division, Naples, Florida
  - Florida Cancer Specialists - North Division, Ocala, Florida
  - Ocala Oncology, Ocala, Florida
  - Florida Cancer Specialists - North Division, Orange City, Florida
  - Florida Cancer Specialists - North Division, Orlando, Florida
  - Florida Cancer Specialists - South Division, Port Charlotte, Florida
  - Florida Cancer Specialists - South Division, Sarasota, Florida
  - Florida Cancer Specialists and Research Institute - North Division, St. Petersburg, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialist - East, Stuart, Florida
  - Florida Cancer Specialists - North Division, Tampa, Florida
  - Florida Cancer Specialists - North Division, Tavares, Florida
  - Florida Cancer Specialists - North Division, Trinity, Florida
  - Florida Cancer Specialists - South Division, Venice, Florida
  - Florida Cancer Specialists - East, Vero Beach, Florida
  - Florida Cancer Specialists - East, Wellington, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Hawaii Cancer Center, Honolulu, Hawaii
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Urology of Indiana, Carmel, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Goshen Health, Goshen, Indiana
  - Our Lady of the Lake, Baton Rouge, Louisiana
  - Pontchartrain, Hammond, Louisiana
  - American Oncology Partners of Maryland PA (Center for Cancer & Blood Disorders), Bethesda, Maryland
  - Frederick Health, Frederick, Maryland
  - Maryland Oncology Hematology, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Central Care Cancer Center, Bolivar, Missouri
  - Lake Regional, Osage Beach, Missouri
  - Mosaic Life Care, Saint Joseph, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - OptumCare Cancer Care-Parent, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Jersey Cancer Care and Blood Disorders, Belleville, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Summit Medical Group - NJ, Florham Park, New Jersey
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - HOACNY, East Syracuse, New York
  - Cayuga Medical Center, Ithaca, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Southeastern Medical Oncology, Goldsboro, North Carolina
  - Sanford Health-Fargo, Fargo, North Dakota
  - Aultman Medical Group, Canton, Ohio
  - TriHealth, Cincinnati, Ohio
  - University of Cincinnati (UC) - Cancer Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Toledo Clinic, Toledo, Ohio
  - Oklahoma State University (OSU) - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialist, Tulsa, Oklahoma
  - Gettysburg-PCSRI, Gettysburg, Pennsylvania
  - Alliance Cancer Specialists, Langhorne, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Cancer Care Associates of York - Parent, York, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Health, Sioux Falls, South Dakota
  - Sarah Cannon and HCA Research Institute, Dickson, Tennessee
  - Sarah Cannon and HCA Research Institute, Franklin, Tennessee
  - Sarah Cannon and HCA Research Institute, Gallatin, Tennessee
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon and HCA Research Institute, Henderson, Tennessee
  - Sarah Cannon and HCA Research Institute, Hermitage, Tennessee
  - Sarah Cannon and HCA Research Institute, Lebanon, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Sarah Cannon and HCA Research Institute, Murfreesboro, Tennessee
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - Sarah Cannon and HCA Research Institute, Shelbyville, Tennessee
  - Sarah Cannon and HCA Research Institute, Smyrna, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology, El Paso, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Arizona Oncology Associates, Irving, Texas
  - Lumi Research, Kingwood, Texas
  - Texas Oncology Central-South, McAllen, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Texas Oncology, Tyler, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Virginia Urology, Richmond, Virginia
  - University of Washington Cancer Consortium, Seattle, Washington
  - Spokane Urology, Spokane, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - ThedaCare, Appleton, Wisconsin
  - Gunderson Health System, La Crosse, Wisconsin
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
- Pan Oncology Trials, LLC, San Juan, Puerto Rico
- South Korea (6):
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No